CLINICAL TRIAL: NCT04422184
Title: Comparative Clinical Evaluation of Three Different Technologies (Novamin, Refix and Refix-k) in Reducing Dental Hypersensitivity in Periodontal Patients
Brief Title: Comparative Clinical Evaluation of Three Different Agents in Reducing Dental Hypersensitivity in Periodontal Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Mariana Ragghianti Zangrando, Assistant professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DHPP60
Record Dates: First submitted 2020-05-29; First posted 2020-06-09 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-05

CONDITIONS: Dentin Hypersensitivity; Periodontal Diseases
Keywords: root exposure; periodontal treatment; desensitizing agents.
MeSH Terms: conditions — Dentin Sensitivity; Periodontal Diseases | interventions — Dentifrices; Potassium Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SEN GROUP (Experimental): Sensodyne Repair and Protect - NOVAMIN technology
  Interventions: Drug: Sensodyne Repair and Protect
- REG GROUP (Experimental): Dentalclean Daily Regenerator - REFIX technology
  Interventions: Drug: Dentalclean Daily Regenerator
- REGK GROUP (Experimental): Dentalclean Daily Regenerator - REFIX technology + potassium citrate
  Interventions: Drug: Dentalclean Daily Regenerator with potassium citrate

INTERVENTIONS:
Drug: Sensodyne Repair and Protect — Dentifricie with NOVAMIN technology
  Other Names: Dentifrice with desensitizing agents
  Arms: SEN GROUP
Drug: Dentalclean Daily Regenerator — Dentifricie with Refix technology
  Other Names: Dentifrice with desensitizing agents
  Arms: REG GROUP
Drug: Dentalclean Daily Regenerator with potassium citrate — Dentifricie with Refix technology+ potassium citrate
  Other Names: Dentifrice with desensitizing agents
  Arms: REGK GROUP

SUMMARY:
The present project will compare the effect of DH reduction using three different dentifrices (Sensodyne Repair and Protect - NOVAMIN technology; Dentalclean Daily Regenerator - REFIX technology; Dentalclean Daily Regenerator - REFIX technology + potassium citrate) in periodontal patients. The evaluation will be in 6 moments: T1 and T2- immediately before and after scaling and root planing (SRP) procedures; T3-after polishing sensitive areas with rubbers cups and the dentifrice determined for each group of patients and T4, 5, 6- After 2, 4 and 8 weeks of SRP. Profissional assessments and patient perception data will be performed.

DETAILED DESCRIPTION:
Periodontal patients may report dentinal hypersensitivity (DH) caused by root surface exposure as part of disease process or as a result of periodontal treatment. Although some studies evaluated DH reduction using desensitizing toothpastes, no specific chemical/physical agent is reported for periodontal patients. Thus, the present project will compare the effect of DH reduction using three different dentifrices (Sensodyne Repair and Protect - NOVAMIN technology; Dentalclean Daily Regenerator - REFIX technology; Dentalclean Daily Regenerator - REFIX technology + potassium citrate) in periodontal patients. This randomized, parallel and blinded clinical trial will be divided into 3 groups (SEN GROUP: Sensodyne; REG GROUP: Regenerator; REGK GROUP: Regenerator + Potassium Citrate) and evaluated at 6 moments: T1 and T2- immediately before and after scaling and root planing (SRP) procedures; T3-after polishing sensitive areas with rubbers cups and the dentifrice determined for each group of patients and T4, 5, 6- After 2, 4 and 8 weeks of SRP. Air blast sensitivity assessments (Schiff scale) and patient perception data on DH will be performed using visual analog scales (VAS). The comparison between treatment groups will be done by paired T-test if normal distribution is observed or Wilcoxon if non-normal distribution. The significance level adopted will be 5% (p <0.05).

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with periodontitis
* 18 to 70 years old
* systemically healthy
* without any allergy to the dentifrices components
* patients who needed scaling and root planing procedures
* patients who had at least 2 teeth with DH (incisors, canines or premolars).

Exclusion Criteria:

* pregnancy
* patients in orthodontic treatment
* patients with oral tumors, caries, fractured teeth, suspected endodontic involvement or excessive mobility;
* patients who used medication that could mask the painful sensation or who had used desensitizing agents in the last 3 months.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2023-05-03 (Actual); Study Completion 2023-05-03 (Actual)

PRIMARY OUTCOMES:
Professional evaluation of Dentin Hypersensitivity | T1- immediately before scaling and root planing procedures (SRP)
  Air blast sensitivity evaluated by an experienced dentist (Schiff scale) Score 0 = Tooth/Subject does not show sensitivity in response to air stimulation; 1 = Tooth/Subject responds to air stimulus, but does not request discontinuation of stimulus; 2 = Tooth/Subject responds to air stimulus, and requests discontinuation or moves from stimulus; 3 = Tooth/Subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Professional evaluation of Dentin Hypersensitivity | T2 - immediately after scaling and root planing procedures (SRP)
  Air blast sensitivity evaluated by an experienced dentist (Schiff scale) Score 0 = Tooth/Subject does not show sensitivity in response to air stimulation; 1 = Tooth/Subject responds to air stimulus, but does not request discontinuation of stimulus; 2 = Tooth/Subject responds to air stimulus, and requests discontinuation or moves from stimulus; 3 = Tooth/Subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Professional evaluation of Dentin Hypersensitivity | T3 - immediately after polishing sensitive areas with rubber cups and the dentifrice determined for each group of patients.
  Air blast sensitivity evaluated by an experienced dentist (Schiff scale) Score 0 = Tooth/Subject does not show sensitivity in response to air stimulation; 1 = Tooth/Subject responds to air stimulus, but does not request discontinuation of stimulus; 2 = Tooth/Subject responds to air stimulus, and requests discontinuation or moves from stimulus; 3 = Tooth/Subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Professional evaluation of Dentin Hypersensitivity | T4 - 2 weeks after SRP.
  Air blast sensitivity evaluated by an experienced dentist (Schiff scale) Score 0 = Tooth/Subject does not show sensitivity in response to air stimulation; 1 = Tooth/Subject responds to air stimulus, but does not request discontinuation of stimulus; 2 = Tooth/Subject responds to air stimulus, and requests discontinuation or moves from stimulus; 3 = Tooth/Subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Professional evaluation of Dentin Hypersensitivity | T5 - 4 weeks after SRP.
  Air blast sensitivity evaluated by an experienced dentist (Schiff scale) Score 0 = Tooth/Subject does not show sensitivity in response to air stimulation; 1 = Tooth/Subject responds to air stimulus, but does not request discontinuation of stimulus; 2 = Tooth/Subject responds to air stimulus, and requests discontinuation or moves from stimulus; 3 = Tooth/Subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Professional evaluation of Dentin Hypersensitivity | T6 - 8 weeks after SRP.
  Air blast sensitivity evaluated by an experienced dentist (Schiff scale) Score 0 = Tooth/Subject does not show sensitivity in response to air stimulation; 1 = Tooth/Subject responds to air stimulus, but does not request discontinuation of stimulus; 2 = Tooth/Subject responds to air stimulus, and requests discontinuation or moves from stimulus; 3 = Tooth/Subject responds to stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.

SECONDARY OUTCOMES:
Patient's perception of DH | T1- immediately before scaling and root planing procedures (SRP)
  Patient's perception of DH was also evaluated with visual analogue scale (VAS), being 0 without any painful sensation and 100 the most painful scenario.
Patient's perception of DH | T2 - immediately after scaling and root planing procedures (SRP)
  Patient's perception of DH was also evaluated with visual analogue scale (VAS), being 0 without any painful sensation and 100 the most painful scenario.
Patient's perception of DH | T3 - immediately after polishing sensitive areas with rubber cups and the dentifrice determined for each group of patients.
  Patient's perception of DH was also evaluated with visual analogue scale (VAS), being 0 without any painful sensation and 100 the most painful scenario.
Patient's perception of DH | T4 - 2 weeks after SRP.
  Patient's perception of DH was also evaluated with visual analogue scale (VAS), being 0 without any painful sensation and 100 the most painful scenario.
Patient's perception of DH | T5 - 4 weeks after SRP.
  Patient's perception of DH was also evaluated with visual analogue scale (VAS), being 0 without any painful sensation and 100 the most painful scenario.
Patient's perception of DH | T6 - 8 weeks after SRP.
  Patient's perception of DH was also evaluated with visual analogue scale (VAS), being 0 without any painful sensation and 100 the most painful scenario.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana S Ragghianti Zangrando, Prof, Principal Investigator — USP
Locations (1):
- Bauru School of Denstistry, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] West NX, Seong J, Davies M. Management of dentine hypersensitivity: efficacy of professionally and self-administered agents. J Clin Periodontol. 2015 Apr;42 Suppl 16:S256-302. doi: 10.1111/jcpe.12336. PMID 25495777
- [Background] Patil SA, Naik BD, Suma R. Evaluation of three different agents for in-office treatment of dentinal hypersensitivity: a controlled clinical study. Indian J Dent Res. 2015 Jan-Feb;26(1):38-42. doi: 10.4103/0970-9290.156796. PMID 25961613